CLINICAL TRIAL: NCT05526586
Title: Twelve Week Safety, Clinical, and Microbiological Efficacy of Experimental Zinc Containing Mouth Rinses
Brief Title: A Twelve Week Study of Prototypes Mouth Rinses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCSORC005014; CCSORC005014 (Other: Johnson & Johnson Consumer Inc.)
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Healthy
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Zero Alcohol Gum Prototype (Experimental): Participants assigned to this group will brush their teeth using a marketed soft bristled toothbrush and Colgate Cavity Protection Toothpaste twice daily and rinse with 20 milliliters (mL) of the Zero Alcohol Gum Prototype Mouth Rinse for 30 seconds, twice a day following brushing on Day 0 under supervision and up to 12 weeks unsupervised at home.
  Interventions: Other: Colgate Cavity Protection Toothpaste; Other: Zero Alcohol Gum Prototype
- Alcohol Gum Prototype (Experimental): Participants assigned to this group will brush their teeth using a marketed soft bristled toothbrush and Colgate Cavity Protection Toothpaste twice daily and rinse with 20 mL of the Alcohol Gum Prototype Mouth Rinse for 30 seconds, twice a day following brushing on Day 0 under supervision and up to 12 weeks unsupervised at home.
  Interventions: Other: Colgate Cavity Protection Toothpaste; Other: Alcohol Gum Prototype
- Listerine Cool Mint Antiseptic Mouthwash (Experimental): Participants assigned to this group will brush their teeth using a marketed soft bristled toothbrush and Colgate Cavity Protection Toothpaste twice daily and rinse with 20 mL of the Listerine Cool Mint Mouth rinse for 30 seconds, twice a day following brushing on Day 0 under supervision and up to 12 weeks unsupervised at home.
  Interventions: Other: Colgate Cavity Protection Toothpaste; Other: Listerine Cool Mint Antiseptic Mouthwash
- Negative Control: 5 percent (%) Hydroalcohol (Active Comparator): Participants assigned to this group will brush their teeth using a marketed soft bristled toothbrush and Colgate Cavity Protection Toothpaste twice daily and rinse with 20 mL of the 5% Hydroalcohol Mouth Rinse for 30 seconds, twice a day following brushing on Day 0 under supervision and up to 12 weeks unsupervised at home.
  Interventions: Other: Colgate Cavity Protection Toothpaste; Other: 5% Hydroalcohol

INTERVENTIONS:
Other: Colgate Cavity Protection Toothpaste — Participants will use Colgate Cavity Protection Toothpaste for brushing teeth twice daily.
Other: Zero Alcohol Gum Prototype — Participants will use 20 mL of Zero Alcohol Gum Prototype Mouth Rinse for 30 seconds after brushing twice daily.
  Arms: Zero Alcohol Gum Prototype
Other: Alcohol Gum Prototype — Participants will use 20 mL of Alcohol Gum Prototype Mouth Rinse for 30 seconds after brushing twice daily.
  Arms: Alcohol Gum Prototype
Other: Listerine Cool Mint Antiseptic Mouthwash — Participants will use 20 mL of Listerine Cool Mint Mouth Rinse for 30 seconds after brushing twice daily.
  Arms: Listerine Cool Mint Antiseptic Mouthwash
Other: 5% Hydroalcohol — Participants will use 20 mL of 5% Hydroalcohol Mouth Rinse for 30 seconds after brushing twice daily.
  Arms: Negative Control: 5 percent (%) Hydroalcohol

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of two essential oil containing experimental mouth rinse formulations and an essential oil containing mouth rinse compared to a hydroalcohol control mouth rinse for the reduction of gingivitis and plaque when used as an adjunct to tooth brushing during a twelve-week product usage period.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and follow the requirements and restrictions of the study (including willingness to use the assigned study products per instructions, availability on scheduled visit dates and likeliness of completing the clinical study) based upon research site personnel's assessment
* Evidence of a personally signed and dated informed consent document indicating the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial
* Able to read and understand the local language (participant is capable of reading the documents)
* Adequate oral hygiene (that is, brush teeth daily and exhibit no signs of oral neglect)
* Adults, 18 years of age and older, in good general and oral health without any known allergy to commercial dental products or cosmetics
* Evidence of being fully vaccinated for coronavirus disease 2019 (COVID-19) (adults 60 years and older)
* Negative pregnancy urine tests (females of child-bearing potential only)
* Females of childbearing potential must be using a medically acceptable method of birth control for at least one month prior to Visit 1 and agree to continue using this method during their participation in the study
* A minimum of 20 natural teeth with scorable facial and lingual surfaces. Teeth that are grossly carious, extensively restored, orthodontically banded, abutments, exhibiting severe generalized cervical and/or enamel abrasion, or third molars will not be included in the tooth count
* A mean gingival index greater than or equal to (>=) 1.95 per the Modified Gingival Index at Baseline
* A mean plaque index >=1.95 per the 6 site Turesky modification of the Quigley-Hein Plaque Index
* Greater than or equal to 10 percent (%) bleeding sites at Baseline
* Absence of significant oral soft tissue pathology, excluding plaque-induced gingivitis, based on a visual examination and at the discretion of the Investigator
* Absence of advanced periodontitis based on a clinical examination and discretion of the dental examiner with probing depths of 4 millimeters (mm) or less except for two sites allowed with a probing depth of 5mm at Baseline
* Absence of fixed or removable orthodontic appliance or removable partial dentures

Exclusion Criteria:

* History of significant adverse effects, including sensitivities or suspected allergies, following use of oral hygiene products such as toothpastes, mouth rinses and red food dye
* Dental prophylaxis within four weeks prior to Baseline visit
* More than two sites that have periodontal pockets depths measuring 5mm or greater in depth
* History of medical conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures
* Use of antibiotics, anti-inflammatory or anticoagulant therapy, phenytoin sodium or diphenylhydantoin, cyclosporin A, immunostimulants/ immunomodulators during the study or within the one month prior to the Baseline exam. Intermittent use of certain anti-inflammatory medication (ibuprofen, Aspirin); oral steroids and calcium channel blockers are acceptable at the discretion of the investigator
* Use of chemotherapeutic anti-plaque/anti-gingivitis products such as triclosan, essential oils, cetylpyridinium chloride, sodium fluoride with CPC, stannous fluoride, zinc or chlorhexidine digluconate containing mouth rinses and toothpastes within the four weeks prior to the Baseline exam
* Known allergy or sensitivity or history of significant adverse effects to any of the investigational product and/or product ingredients (or other ingredients in the products)
* Consumption of probiotic drinks/supplements within one week prior to Screening/Baseline
* Self-reported pregnancy or lactation (this criterion is due to oral tissue changes related to pregnancy and nursing which can affect interpretation of study results)
* Self-reported smokeless tobacco user including snuff, chewing tobacco, vaping and e-cigarette usage
* Males with a pregnant partner or a partner who is currently trying to become pregnant
* Suspected alcohol or substance abuse (example, amphetamines, benzodiazepines, cocaine, marijuana, opiates)
* Significant medical or oral condition which may interfere with a subject's participation in the study, including cancer, chronic kidney disease, COPD (chronic obstructive pulmonary disease), immunocompromised state (weakened immune system) from solid organ transplant, serious heart conditions, (such as heart failure, coronary artery disease, or cardiomyopathies) Sickle cell disease, Type 2 diabetes mellitus at the discretion of the Investigator
* Participation in any clinical trial within 30 days of Screening visit
* Diagnosed Temporo-mandibular joint dysfunction/disorder
* Subjects who wear bruxing devices, dental aligners, retainers
* Subjects who were previously screened and ineligible or were randomized to receive investigational product
* Subjects who are related to those persons involved directly or indirectly with the conduct of this study (that is, principal investigator, sub-investigators, study coordinators, other site personnel, employees of Johnson & Johnson subsidiaries, contractors of Johnson & Johnson, and the families of each)
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study
* COVID-19 restrictions: Participants who fail to meet the criteria of the site's screening consent for Preventing Infection in the site's COVID-19 consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2022-08-31 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Whole-mouth Mean Modified Gingival Index (MGI) Score After 12 Weeks of Product use | After 12 weeks
  Gingivitis will be assessed by the MGI on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth: 0 (Normal [absence of inflammation]), 1 (Mild inflammation [slight change in color, little change in texture] of any portion of the entire gingival unit); 2 (Mild inflammation of the entire gingival unit); 3 (Moderate inflammation [moderate glazing, redness, edema, and/or hypertrophy] of the gingival unit); 4 (Severe inflammation [marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration] of the gingival unit).
Whole-mouth Mean Plaque Index (TPI) Score After 12 Weeks of Product use | After 12 weeks
  Plaque area will be scored by the Turesky modification of the Quigley-Hein Plaque Index, on 6 surfaces (distobuccal, midbuccal and mesiobuccal, distolingual, midlingual and mesiolingual) of all scorable teeth, following disclosing: 0 (No Plaque); 1 (Separate flecks or discontinuous band of plaque around the gingival (cervical) margin); 2 (Thin (up to 1 millimeter [mm]), continuous band of plaque at the gingival margin); 3 (Band of plaque wider than 1mm but less than 1/3 of the surface); 4 (Plaque covering 1/3 or more, but less than 2/3 of the surface); 5 (Plaque covering 2/3 or more of the surface).

SECONDARY OUTCOMES:
Whole-mouth Mean TPI Score After 1 and 4 Weeks of Product use | After Weeks 1 and 4
  Plaque area will be scored by the Turesky modification of the Quigley-Hein Plaque Index, on 6 surfaces (distobuccal, midbuccal and mesiobuccal, distolingual, midlingual and mesiolingual) of all scorable teeth, following disclosing: 0 (No Plaque); 1 (Separate flecks or discontinuous band of plaque around the gingival (cervical) margin); 2 (Thin [up to 1 mm], continuous band of plaque at the gingival margin); 3 (Band of plaque wider than 1mm but less than 1/3 of the surface); 4 (Plaque covering 1/3 or more, but less than 2/3 of the surface); 5 (Plaque covering 2/3 or more of the surface).
Whole-mouth Mean MGI Score After 1 and 4 Weeks of Product Use | After 1 and 4 weeks
  Gingivitis will be assessed by the MGI on the buccal and lingual marginal gingivae and interdental papillae of all scorable teeth: 0 (Normal [absence of inflammation]), 1 (Mild inflammation [slight change in color, little change in texture] of any portion of the entire gingival unit); 2 (Mild inflammation of the entire gingival unit); 3 (Moderate inflammation [moderate glazing, redness, edema, and/or hypertrophy] of the gingival unit); 4 (Severe inflammation [marked redness and edema/hypertrophy, spontaneous bleeding, or ulceration] of the gingival unit).
Whole-Mouth Mean Expanded Gingival Bleeding Index (EBI) Score at 1, 4 and 12 Weeks of Product use | Weeks 1, 4 and 12
  Bleeding will be assessed according to the EBI, 168 Sites. A periodontal probe with a 0.5 mm diameter tip will be inserted into the gingival crevice and swept from distal to mesial around the tooth at an angle of approximately 60 degrees, while in contact with the sulcular epithelium. Each of 6 gingival areas (distobuccal, mid-buccal, mesiobuccal, distolingual, mid-lingual, and mesiolingual) around each tooth will be assessed. After approximately 30 seconds, bleeding at each gingival unit will be recorded according to the following scale: 0 (Absence of bleeding after 30 seconds); 1 (Bleeding after 30 seconds); 2 (Immediate bleeding).
Percentage of Bleeding Sites, Based on the EBI Score at 1, 4, and 12 Weeks of Product use | After 1, 4, and Week 12
  Percentage of bleeding sites will be calculated by taking the total number of sites with bleeding score greater than 0 divided by the total number of sites assessed for each participant. Bleeding will be assessed according to the Expanded Gingival Bleeding Index, 168 Sites. A periodontal probe with a 0.5 mm diameter tip will be inserted into the gingival crevice and swept from distal to mesial around the tooth at an angle of approximately 60 degrees, while in contact with the sulcular epithelium. Each of 6 gingival areas (distobuccal, mid-buccal, mesiobuccal, distolingual, mid-lingual, and mesiolingual) around each tooth will be assessed. After approximately 30 seconds, bleeding at each gingival unit will be recorded according to the following scale: 0 (Absence of bleeding after 30 seconds); 1 (Bleeding after 30 seconds); 2 (Immediate bleeding).
Whole Mouth Bleeding on Probing Depth at 12 Week | At Week 12
  Whole mouth bleeding on probing depth at 12 week will be reported.
Number of Distinct Bacterial Species | At Baseline and 1, 4, and 12 weeks
  The number of distinct bacterial species identified on supragingival plaque using microbiome profiling will be reported at baseline, 1 week, 4 weeks and 12 weeks.
Shannon-weaver Diversity Index | At Baseline and 1, 4, and 12 weeks
  The Shannon-Weaver diversity index will be reported for supragingival plaque assessment.
Total Species Microbial Load | At Baseline and 1, 4, and 12 weeks
  The total species microbial load will be reported for supragingival plaque assessment.
Categorical Species Microbial Load | At Baseline and 1, 4, and 12 weeks
  The categorical species microbial load will be reported for supragingival plaque assessment.
Changes in Microbiome Composition by Sample Clustering Analysis | At Baseline and 1, 4, and 12 weeks
  Clustering analysis in microbiome profiling is a multidimensional reduction analysis for the assessment of microbiome composition shift.
Number of Live Bacterial Counts Expressed in Log10 | At Baseline and After 12 weeks
  The number of live bacterial counts (expressed in log10) on supragingival and subgingival plaque will be reported at baseline and 12 weeks using viability quantitative polymerase chain reaction (qPCR) targeting total bacteria, Fusobacterium nucleatum, Porphyromonas gingivalis and Actinomyces oris.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Milleman, DDS, Principal Investigator — Salus Research, Inc.
Locations (1):
- Salus Research, Inc., Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu

REFERENCES:
- See also: Twelve Week Safety, Clinical, and Microbiological Efficacy of Experimental Zinc Containing Mouth Rinses — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CCSORC005014&attachmentIdentifier=affa4e64-746a-4874-801f-d9568281dff7&fileName=CCSORC005014___CSR_Synopsis__Flat.pdf&versionIdentifier=